CLINICAL TRIAL: NCT01686178
Title: Countering Young Adult Tobacco Marketing in Bars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01CA154240-05 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Smoking Cessation
Keywords: Smoking; Smoking Cessation; Tobacco Use Cessation; Social Networks; Social Control, Informal
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-smoking social marketing campaign (Experimental): In prior research, a high risk subpopulation of young adults was identified in San Diego, CA: the "hipster" subculture. We developed a yearlong pilot social branding intervention to decrease smoking among this group, using social events and social leaders to promote a strong nonsmoking lifestyle. The intervention rationale is based on utilizing industry market research tools to define the target audience and directly countering tobacco industry lifestyle marketing strategies. We now propose to extend this intervention to three other cities (tailoring the intervention to a high-risk subpopulation of young adults in each city) and evaluate it in a multicenter quasi-experimental controlled trial.
  Interventions: Behavioral: Anti-smoking social marketing campaign
- Control (No Intervention): Survey research data will be collected in control cities with the same schedule as data collection in the cities where the intervention is taking place.

INTERVENTIONS:
Behavioral: Anti-smoking social marketing campaign — We will utilize industry market research tools to define the target audience (segment of community with high smoking prevalence and high social influence) and directly counter tobacco industry lifestyle marketing strategies through local promotion of a smokefree brand and branded bar and club events.
  Arms: Anti-smoking social marketing campaign

SUMMARY:
The goal of the study is to implement and evaluate interventions to decrease smoking among young adults attending bars and nightclubs. It is believed that the proportion of young adult current smokers during and after the intervention will be significantly less than the proportion of young adult smokers before the intervention in each of the study cities.

ELIGIBILITY:
Inclusion Criteria:

* Participants are healthy volunteers 18-26 years old currently living in San Diego, Portland, Albuquerque, Oklahoma, San Francisco/Bay Area, Nashville, Tucson, or Los Angeles who attend bars or nightclubs
* Able to read, speak, and understand English
* NOTE: PARTICIPANTS CAN ONLY TAKE PART IN THE STUDY BY ENCOUNTERING STUDY SURVEY TEAMS OUT AT BARS OR NIGHTCLUBS IN ONE OF THE STUDY CITIES LISTED ABOVE. PARTICIPANTS CANNOT SIGN UP FOR THE STUDY BY CALLING OR EMAILING.

Exclusion Criteria:

* Out of age range (18-26 years old)
* Not living in San Diego, Portland, Albuquerque, Oklahoma, San Francisco/Bay Area, Nashville, Tucson, Los Angeles or New York City, or currently attending college outside of the target cities.
* Unable to read, speak, or understand English.
* Unwillingness or inability to participate or give informed consent.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17422 (Actual)
Dates: Start 2012-09; Primary Completion 2017-07-02 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
Self-Reported Tobacco Smoking in past 30 days | Between baseline and follow-up at 1,2, & 3 years post-baseline
  The main outcome measure for this analysis will be the proportion of current smoking, defined as self-reported smoking on one or more of the past 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela M Ling, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Ling PM, Glantz SA. Using tobacco-industry marketing research to design more effective tobacco-control campaigns. JAMA. 2002 Jun 12;287(22):2983-9. doi: 10.1001/jama.287.22.2983. PMID 12052128
- [Derived] Ling PM, Lisha NE, Neilands TB, Jordan JW. Join the Commune: A Controlled Study of Social Branding Influencers to Decrease Smoking Among Young Adult Hipsters. Am J Health Promot. 2020 Sep;34(7):754-761. doi: 10.1177/0890117120904917. Epub 2020 Feb 20. PMID 32077305
- [Derived] Lisha NE, Jordan JW, Ling PM. Peer crowd affiliation as a segmentation tool for young adult tobacco use. Tob Control. 2016 Oct;25(Suppl 1):i83-i89. doi: 10.1136/tobaccocontrol-2016-053086. PMID 27697952